CLINICAL TRIAL: NCT03321513
Title: Randomized Trial of Intravitreous Aflibercept Versus Intravitreous Bevacizumab + Deferred Aflibercept for Treatment of Central-Involved Diabetic Macular Edema
Brief Title: DRCR.Net Aflibercept vs. Bevacizumab + Deferred Aflibercept for the Treatment of CI-DME
Acronym: DRCR AC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AC
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; anti-vascular endothelial growth factor
MeSH Terms: interventions — aflibercept; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept Group (Active Comparator): 2.0 mg intravitreous aflibercept
  Interventions: Drug: intravitreous aflibercept
- Bevacizumab + Deferred Aflibercept Group (Experimental): 1.25 mg intravitreous bevacizumab + deferred intravitreous 2.0 mg aflibercept if eye meets switch criteria
  Interventions: Drug: intravitreous aflibercept; Drug: Bevacizumab + Deferred Aflibercept Group

INTERVENTIONS:
Drug: intravitreous aflibercept — Intravitreous aflibercept injection is made by Regeneron Pharmaceuticals, Inc. and is approved by the FDA for the treatment of neovascular age-related macular degeneration, macular edema due to central retinal vein occlusion, macular edema due to branch retinal vein occlusion, diabetic macular edema, and diabetic retinopathy in eyes with diabetic macular edema.
  Study eyes assigned to receive aflibercept will receive a dose of 2.0 mg in 0.05 cc. Aflibercept will be obtained commercially by the clinical site. The physical, chemical, and pharmaceutical properties and formulation of aflibercept are provided in the Package Insert.
  Intravitreous Injection Technique The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using sterile technique
  Other Names: Eylea
Drug: Bevacizumab + Deferred Aflibercept Group — Bevacizumab is made by Genentech, Inc. and is approved by the FDA for the treatment of metastatic colorectal cancer as well as the treatment of non-squamous non-small cell lung cancer, glioblastoma, and metastatic renal cell carcinoma.
  Study eyes assigned to receive bevacizumab will receive a dose of 1.25 mg provided by a single compounding pharmacy identified by the Network and distributed by the Network. The volume of the injections will be 0.05 cc.
  Intravitreous injection technique: The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using a sterile technique.
  Other Names: Avastin
  Arms: Bevacizumab + Deferred Aflibercept Group

SUMMARY:
Both aflibercept and bevacizumab have been shown to improve vision in eyes with DME. In eyes with DME and at least moderate vision loss, both aflibercept and bevacizumab were also shown to be successful in many eyes. However, aflibercept was shown to be more effective at improving vision, on average, at 1 year and at 2 years. Due to the large cost difference between the two drugs, many clinicians and patients are choosing to initiate treatment with bevacizumab and then switch to aflibercept depending on the eye's response to bevacizumab treatment. However, there is no scientific evidence that this treatment strategy is as effective at improving vision as initiating treatment with aflibercept. Patients and clinicians do not know if this approach ultimately has deleterious effects on visual acuity. If starting with aflibercept is not better than starting with bevacizumab and switching to aflibercept if needed, the potential cost savings to future patients and the health care system would be substantial. However, if starting with aflibercept is better, then patients, clinicians, and health care providers can make informed decisions for how to best treat patients with DME and at least moderate vision loss.

Study Objectives To compare the efficacy of intravitreous aflibercept with intravitreous bevacizumab + deferred aflibercept if needed in eyes with CI DME and moderate vision loss

ELIGIBILITY:
Participant-level Criteria Inclusion

To be eligible, the following inclusion criteria must be met:

1. Age ≥ 18 years • Individuals <18 years old are not being included because DME is so rare in this age group that the diagnosis of DME may be questionable.
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   * Any one of the following will be considered to be sufficient evidence that diabetes is present:

   Current regular use of insulin for the treatment of diabetes Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes Documented diabetes by American Diabetes Association and/or World Health Organization criteria
3. At least one eye meets the study eye criteria listed.
4. Able and willing to provide informed consent.

   Exclusion

   An individual is not eligible if any of the following exclusion criteria are present:
5. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
6. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).

   * Individuals in poor glycemic control who, within the last four months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next four months should not be enrolled.
7. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied at the time of study entry.

   • Note: study participants cannot receive another investigational drug while participating in the study.
8. Known allergy to any component of the study drug or any drug used in the injection prep (including povidone iodine prep).
9. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).

   • If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
10. Systemic anti-VEGF or pro-VEGF treatment within four months prior to randomization or anticipated use during the study.

    • These drugs cannot be used during the study.
11. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 24 months.

    • Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
12. Individual is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next two years.

Study Eye Criteria The study participant must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below.

Study participants can have two study eyes only if both eyes are eligible at the time of randomization. For study participants with two eligible eyes, the logistical complexities of the protocol must be considered for each individual prior to randomizing both eyes.

The eligibility criteria for a study eye are as follows:

Inclusion

1. Best corrected Electronic-Early Treatment Diabetic Retinopathy Study visual acuity letter score < 69 (i.e., 20/50 or worse) and ≥ 24 (i.e., 20/320 or better) within eight days of randomization.
2. On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula.
3. Diabetic macular edema present on optical coherence tomography (OCT) within eight days of randomization

   * Zeiss Cirrus central subfield: ≥ 290µm in women or ≥ 305µm in men
   * Heidelberg Spectralis central subfield: ≥ 305µm in women or ≥ 320µm in men
   * Investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality
4. Media clarity, pupillary dilation, and individual cooperation sufficient for adequate fundus photographs.

   Exclusions

   The following exclusions apply to the study eye only (i.e., they may be present for the nonstudy eye):
5. Macular edema is considered to be due to a cause other than diabetic macular edema.

   • An eye should not be considered eligible if: (1) the macular edema is considered to be related to ocular surgery such as cataract extraction or (2) clinical exam and/or OCT suggest that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are the primary cause of the macular edema.
6. An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
7. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
8. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
9. History of an anti-vascular endothelial growth factor (anti-VEGF) treatment for diabetic macular edema (DME) in the past 12 months or history of any other treatment for DME at any time in the past four months (such as focal/grid macular photocoagulation, intravitreous or peribulbar corticosteroids).

   • Enrollment will be limited to a maximum of 25% of the planned sample size with any history of anti-VEGF treatment for DME. Once this number of eyes has been enrolled, any history of anti-VEGF treatment for DME will be an exclusion criterion.
10. History of pan-retinal photocoagulation within four months prior to randomization or anticipated need for pan-retinal photocoagulation in the six months following randomization.
11. History of anti-VEGF treatment for a disease other than DME in the past 12 months.
12. History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior four months or anticipated within the next six months following randomization.
13. History of YAG capsulotomy performed within two months prior to randomization.
14. Aphakia.
15. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.
16. Evidence of uncontrolled glaucoma. • Intraocular pressure must be <30, with no more than one topical glaucoma medication, and no documented glaucomatous field loss for the eye to be eligible

Note, combination therapies are considered more than one medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Retinal Diagnostic Center, Campbell, California
  - Macula & Retina Institute, Glendale, California
  - Loma Linda University Health Care, Department of Ophthalmology, Loma Linda, California
  - East Bay Retina Consultants, Inc, Oakland, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Retina Institute-Jacksonville, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Retina Macula Specialists of Miami, Miami, Florida
  - Central Florida Retina, Orlando, Florida
  - Florida Retina Institute, Orlando, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Retina Specialists of Tampa, Wesley Chapel, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Illinois Retina Associates, S.C., Oak Park, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - The Retina Institute, St Louis, Missouri
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - MaculaCare, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Western Carolina Clinical Research, LLC, Asheville, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Cascade Medical Research Institute, LLC, Springfield, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Retinavitreous Associates, dba; Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina Center of Texas, Grapevine, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Spokane Eye Clinic, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jhaveri CD, Glassman AR, Ferris FL 3rd, Liu D, Maguire MG, Allen JB, Baker CW, Browning D, Cunningham MA, Friedman SM, Jampol LM, Marcus DM, Martin DF, Preston CM, Stockdale CR, Sun JK; DRCR Retina Network. Aflibercept Monotherapy or Bevacizumab First for Diabetic Macular Edema. N Engl J Med. 2022 Aug 25;387(8):692-703. doi: 10.1056/NEJMoa2204225. Epub 2022 Jul 14. PMID 35833805

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with both eyes enrolled had one eye in each group (N = 42). Participants could have had 1 (unilateral) or each eye (bilateral) assigned to each group. "Unilateral: "Aflibercept- Monotherapy Group" only (116 participants), "Bevacizumab-First Group" only (112 participants); Bilateral: 42 participants
Units Other Than Participants: Eyes
Groups:
- Aflibercept- Monotherapy Group: 2.0 mg intravitreous aflibercept
  intravitreous aflibercept: Intravitreous aflibercept injection is made by Regeneron Pharmaceuticals, Inc. and is approved by the FDA for the treatment of neovascular age-related macular degeneration, macular edema due to central retinal vein occlusion, macular edema due to branch retinal vein occlusion, diabetic macular edema, and diabetic retinopathy in eyes with diabetic macular edema.
  Study eyes assigned to receive aflibercept will receive a dose of 2.0 mg in 0.05 cc. Aflibercept will be obtained commercially by the clinical site. The physical, chemical, and pharmaceutical properties and formulation of aflibercept are provided in the Package Insert.
  Intravitreous Injection Technique The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using sterile technique
- Bevacizumab-First Group: 1.25 mg intravitreous bevacizumab + deferred intravitreous 2.0 mg aflibercept if eye meets switch criteria
  Bevacizumab + Deferred Aflibercept Group: Bevacizumab is made by Genentech, Inc. and is approved by the FDA for the treatment of metastatic colorectal cancer as well as the treatment of non-squamous non-small cell lung cancer, glioblastoma, and metastatic renal cell carcinoma.
  Study eyes assigned to receive bevacizumab will receive a dose of 1.25 mg provided by a single compounding pharmacy identified by the Network and distributed by the Network. The volume of the injections will be 0.05 cc.
  Intravitreous injection technique: The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using a sterile technique.
Period: Overall Study
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Started | 158; 158 Eyes (There were 42 participants with both eyes enrolled, one in each group.) | 154; 154 Eyes (There were 42 participants with both eyes enrolled, one in each group.)
Completed | 132; 132 Eyes | 128; 128 Eyes
Not Completed | 26; 26 Eyes | 26; 26 Eyes
Not completed — Death | 11 | 5
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Lost to Follow-up | 10 | 11

BASELINE CHARACTERISTICS:
Population: Units in Eyes
Units Other Than Participants: Eyes
Groups:
- Bevacizumab-First Group: 1.25 mg intravitreous bevacizumab + deferred intravitreous 2.0 mg aflibercept if eye meets switch criteria.
  1.25 mg intravitreous bevacizumab was administered at randomization and thereafter according to the prespecified retreatment protocol. Beginning at 12 weeks, and only if protocol-specified criteria were met, eyes in this group stopped bevacizumab therapy and started aflibercept therapy. Bevacizumab + Deferred Aflibercept Group: Bevacizumab is made by Genentech, Inc. and is approved by the FDA for the treatment of metastatic colorectal cancer as well as the treatment of non-squamous non-small cell lung cancer, glioblastoma, and metastatic renal cell carcinoma.
  Study eyes assigned to receive bevacizumab will receive a dose of 1.25 mg provided by a single compounding pharmacy identified by the Network and distributed by the Network. The volume of the injections will be 0.05 cc.
  Intravitreous injection technique: The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using a sterile technique.
- Total: Total of all reporting groups
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group | Total
Number analyzed (Participants) | 158 | 154 | 270
Number analyzed (Eyes) | 158 | 154 | 312
Age, Customized [Median (Inter-Quartile Range); unit: years] — Population: 84 eyes were enrolled with from 42 participants with two study eyes (i.e., one eye in each treatment group).
  years
    age | 60 [55 to 66] | 61 [54 to 67] | 61 [54 to 66]
Sex/Gender, Customized [Count of Units; unit: Eyes]
  Women | 76 | 74 | 150
  Male | 82 | 80 | 162
Race/Ethnicity, Customized [Count of Units; unit: Eyes] — Population: 84 eyes were enrolled with from 42 participants with two study eyes (i.e., one eye in each treatment group).
  Eyes
    White | 82 | 83 | 165
    Black or African American | 32 | 26 | 58
    Hispanic or Latino | 39 | 41 | 80
    Asian | 2 | 2 | 4
    Native Hawaiian or other Pacific Islander | 1 | 1 | 2
    Multiple | 1 | 1 | 2
    Unknown or not reported | 1 | 0 | 1
Type of diabetes [Count of Units; unit: Eyes] — Population: 84 eyes were enrolled with from 42 participants with two study eyes (i.e., one eye in each treatment group).
  Eyes
    Type 1 | 7 | 8 | 15
    Type 2 | 151 | 146 | 297
Duration of diabetes [Median (Inter-Quartile Range); unit: years] | 15 [9 to 21] | 14 [5 to 21] | 15 [7 to 21]
Glycated hemoglobin [Median (Inter-Quartile Range); unit: Hemoglobin A1c percentage] — Population: Data on the glycated hemoglobin level were unavailable for 10 eyes in each trial group.
  Hemoglobin A1c percentage
    number analyzed (Participants) | 148 | 144 | 255
    number analyzed (Eyes) | 148 | 144 | 292
    (all) | 8.0 [7.2 to 9.4] | 8.0 [6.8 to 9.4] | 8.0 [6.9 to 9.4]
Visual acuity letter score [Median (Inter-Quartile Range); unit: units on a scale] — Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity. Population: 84 eyes were enrolled with from 42 participants with two study eyes (i.e., one eye in each treatment group).
  units on a scale | 61 [54 to 65] | 60 [51 to 65] | 60 [52 to 65]
Central subfield thickness [Median (Inter-Quartile Range); unit: Microns] — Measurements made on the Cirrus optical coherence tomography device were converted to equivalent scores as would be assessed on the Spectralis optical coherence tomography device with the use of the following formula: Spectralis score = 40.78 + 0.95 × Cirrus score. Population: Data were unavailable for two eyes in the aflibercept-monotherapy group; a optical coherence tomography reading center confirmed the presence of diabetic macular edema in these eyes.
  84 eyes were enrolled with from 42 participants with two study eyes (i.e., one eye in each treatment group).
  Microns
    number analyzed (Participants) | 156 | 154 | 269
    number analyzed (Eyes) | 156 | 154 | 310
    (all) | 478 [401 to 579] | 496 [407 to 628] | 488 [404 to 616]
Diabetic retinopathy severity scale [Count of Units; unit: Eyes] — Severity levels include 12 discrete steps ranging from 10 to 85, with higher levels indicating greater severity. Level was based on assessment by the reading center. Population: Data were not available for one eye in the bevacizumab-first group. Eyes could not be graded for seven eyes in the aflibercept-monotherapy group and for six eyes in the bevacizumab-first group. Percentages are based on the numbers of eyes with gradable severity of diabetic retinopathy at baseline.
  84 eyes were enrolled with from 42 participants with two study eyes (i.e., one eye in each treatment group).
  Eyes
    number analyzed (Participants) | 151 | 147 | 258
    number analyzed (Eyes) | 151 | 147 | 298
    Diabetic retinopathy absent or questionable; levels 10, 12, 14, or 15 | 0 | 1 | 1
    Microaneurysms only; level 20 | 0 | 2 | 2
    Mild-to-moderate nonproliferative diabetic retinopathy; level 35 or 43 | 58 | 42 | 100
    Moderately severe to severe nonproliferative diabetic retinopathy; level 47 or 53 | 72 | 79 | 151
    Mild-to-moderate proliferative diabetic retinopathy; level 61 or 65 | 15 | 16 | 31
    High-risk proliferative diabetic retinopathy; level 71 or 75 | 6 | 7 | 13
    Advanced Proliferative diabetic retinopathy Level 81 or 85 | 0 | 0 | 0
Previous anti-VEGF treatment for diabetic macular edema [Number; unit: Eyes] — anti-VEGF = vascular endothelial growth factor.
  Eyes | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity
Description: Area under the curve mean change in the electronic early treatment diabetic retinopathy study visual acuity. Visual acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study visual-acuity test on a scale from 100 letters (Snellen equivalent, 20/10) to 0 letters (Snellen equivalent, <20/800), with higher scores indicating better vision. The data presented are the best-corrected visual acuity in the study eye after protocol-defined refraction. The primary outcome was the time-averaged change in the visual-acuity letter score over a period of 104 weeks. The score was derived by calculating the area under the curve (AUC) over the 104-week period for the change in visual acuity from baseline and dividing by the length of follow-up.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 132 | 128
Number analyzed (Eyes) | 132 | 128
Letter Score | 15 (8.5) | 14 (8.8)

2. Secondary Outcome: Change in Visual Acuity From Baseline
Description: Visual acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study visual-acuity test on a scale from 100 letters (Snellen equivalent, 20/10) to 0 letters (Snellen equivalent, <20/800), with higher scores indicating better vision.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 132 | 128
Number analyzed (Eyes) | 132 | 128
Letter Score | 14.7 (14.5) | 15.9 (12.4)

3. Secondary Outcome: Increase in E-ETDRS Visual Acuity Letter Score
Description: Visual acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual-acuity test on a scale from 100 letters (Snellen equivalent, 20/10) to 0 letters (Snellen equivalent, <20/800), with higher scores indicating better vision.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 132 | 128
Number analyzed (Eyes) | 132 | 128
Eyes
  15 or more letters | 70 | 74
  10 or more letters | 101 | 98

4. Secondary Outcome: Decrease in E-ETDRS Visual Acuity Letter Score
Description: as for outcome 2
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 132 | 128
Number analyzed (Eyes) | 132 | 128
Eyes
  15 or more letters | 9 | 5
  10 or more letters | 8 | 4

5. Secondary Outcome: Visual Acuity
Description: as for outcome 2
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 132 | 128
Number analyzed (Eyes) | 132 | 128
Eyes
  20/20 or better | 29 | 28
  20/40 or worse | 96 | 95
  20/200 or worse | 6 | 2

6. Secondary Outcome: Optical Coherence Tomography Central Subfield Thickness Change From Baseline
Description: Measurements made on the Cirrus device were converted to equivalent scores as would be assessed on the Spectralis device with the use of the following formula: Spectralis score = 40.78 + 0.95 × Cirrus score.
Time Frame: 2 years
Population: The analysis included only eyes for which baseline data on the central subfield thickness were available.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 126 | 127
Number analyzed (Eyes) | 126 | 127
microns | -192 (143) | -198 (160)

7. Secondary Outcome: Optical Coherence Tomography Central Subfield Thickness Below the Sex-specific Threshold for Central-involved Diabetic Macular Edema
Description: Optical coherence tomography (OCT) central subfield thickness equivalents for measurements obtained on Spectral domain OCT machines were 320 μm for men and 305 μm for women on the Spectralis device (Heidelberg) and were 305 μm and 290 μm, respectively on the Cirrus OCT measurement device (Zeiss).
Time Frame: 2 years
Population: The analysis included only eyes for which baseline data on the central subfield thickness were available.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 126 | 127
Number analyzed (Eyes) | 126 | 127
Eyes | 76 | 70

8. Secondary Outcome: Number of Visits
Time Frame: 2 years
Population: This analysis was limited to patients with one study eye who completed 2 years of follow-up.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 98 | 94
visits | 22.0 (3.6) | 22.5 (3.4)

9. Secondary Outcome: Number of Injections
Description: All study injections were counted, including aflibercept injections received among eyes in the bevacizumab first group.
Time Frame: 2 years
Population: Limited to eyes that completed the 2-year visit or any later common visit.
Measure: Mean (Standard Deviation); unit: injections
Units Other Than Participants: Eyes
Arm/Group | Aflibercept- Monotherapy Group | Bevacizumab-First Group
Number analyzed (Participants) | 132 | 128
Number analyzed (Eyes) | 132 | 128
injections | 14.6 (4.1) | 16.1 (4.1)

10. Secondary Outcome: Number of Eyes in the Bevacizumab-first Group Meeting the Switching Criteria
Time Frame: Baseline to 12 weeks
Population: Eyes that did not meet the switch criteria were censored at the last completed visit
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bevacizumab-First Group
Number analyzed (Participants) | 154
Number analyzed (Eyes) | 154
Eyes | 16

11. Secondary Outcome: Number of Eyes in the Bevacizumab-first Group Meeting the Switching Criteria
Time Frame: Baseline to 24 weeks
Population: Eyes that did not meet the switch criteria were censored at the last completed visit
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bevacizumab-First Group
Number analyzed (Participants) | 154
Number analyzed (Eyes) | 154
Eyes | 57

12. Secondary Outcome: Number of Eyes in the Bevacizumab-first Group Meeting the Switching Criteria
Time Frame: Baseline to 52 weeks
Population: Eyes that did not meet the switch criteria were censored at the last completed visit
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bevacizumab-First Group
Number analyzed (Participants) | 154
Number analyzed (Eyes) | 154
Eyes | 88

13. Secondary Outcome: Number of Eyes in the Bevacizumab-first Group Meeting the Switching Criteria
Time Frame: Baseline to 104 weeks
Population: Eyes that did not meet the switch criteria were censored at the last completed visit
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bevacizumab-First Group
Number analyzed (Participants) | 154
Number analyzed (Eyes) | 154
Eyes | 100

ADVERSE EVENTS:
Time Frame: 2 Years
Description: To get the total number of participant/eyes in each treatment group add the unilateral and bilateral participants together:
  Unilateral Aflibercept monotherapy = 116 Total Aflibercept monotherapy = unilateral Aflibercept monotherapy + bilateral = 116 + 42 = 158 Unilateral Bevacizumab first = 112 total Bevacizumab first = unilateral Bevacizumab first + bilateral = 112 + 42 = 154.
Groups:
- Unilateral Aflibercept- Monotherapy Group: 2.0 mg intravitreous aflibercept
  intravitreous aflibercept: Intravitreous aflibercept injection is made by Regeneron Pharmaceuticals, Inc. and is approved by the FDA for the treatment of neovascular age-related macular degeneration, macular edema due to central retinal vein occlusion, macular edema due to branch retinal vein occlusion, diabetic macular edema, and diabetic retinopathy in eyes with diabetic macular edema.
  Study eyes assigned to receive aflibercept will receive a dose of 2.0 mg in 0.05 cc. Aflibercept will be obtained commercially by the clinical site. The physical, chemical, and pharmaceutical properties and formulation of aflibercept are provided in the Package Insert.
  Intravitreous Injection Technique The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using sterile technique.
- Unilateral Bevacizumab-First Group: 1.25 mg intravitreous bevacizumab + deferred intravitreous 2.0 mg aflibercept if eye meets switch criteria
  Bevacizumab + Deferred Aflibercept Group: Bevacizumab is made by Genentech, Inc. and is approved by the FDA for the treatment of metastatic colorectal cancer as well as the treatment of non-squamous non-small cell lung cancer, glioblastoma, and metastatic renal cell carcinoma.
  Study eyes assigned to receive bevacizumab will receive a dose of 1.25 mg provided by a single compounding pharmacy identified by the Network and distributed by the Network. The volume of the injections will be 0.05 cc.
  Intravitreous injection technique: The injection is preceded by a povidone iodine prep of the conjunctiva. In general, topical antibiotics in the pre-, peri-, or post-injection period should not be used.
  The injection will be performed using a sterile technique. For participants who switched from Bevacizumab to Aflibercept, all randomized eyes are included in the safety analysis and analyzed according to treatment assignment at randomization, regardless of the treatment actually received.
- Bilateral Participants: Participants with one eye enrolled in each arm of the study. For participants who switched from Bevacizumab to Aflibercept, all randomized eyes are included in the safety analysis and analyzed according to treatment assignment at randomization, regardless of the treatment actually received.
  Ocular adverse events specific to each treatment are reported as footnotes.
Arm/Group | Unilateral Aflibercept- Monotherapy Group | Unilateral Bevacizumab-First Group | Bilateral Participants
All-Cause Mortality (participants affected / at risk) | 10/116 | 4/112 | 3/42
Serious Adverse Events (participants affected / at risk) | 61/116 | 42/112 | 18/42
Other Adverse Events (participants affected / at risk) | 100/116 | 94/112 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unilateral Aflibercept- Monotherapy Group (N=116) | Unilateral Bevacizumab-First Group (N=112) | Bilateral Participants (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Anemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Enlargement of lymph nodes (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
AFib (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital heart disease NOS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 9 (11) | 1 (1) | 4 (4)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Worsening of diabetes (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Double vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Bevacizumab-First Group.
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Penetrating eye injury (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (13) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gastro intestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach virus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 2 (2) | 0 (0)
Death (General disorders) | 4 (4) | 0 (0) | 1 (1)
General Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
E. coli infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Foot infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural hematoma (traumatic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Blood sugar decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased hemoglobin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased white cell count (Investigations) | 1 (1) | 0 (0) | 0 (0)
Elevated liver enzymes (Investigations) | 1 (1) | 0 (0) | 0 (0)
Potassium high (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Water retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Broken bones (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fractured ethmoid (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fractured maxilla (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Necrotizing fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Brain tumor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Consciousness loss (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fainting (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness facial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Shakiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental state abnormal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic renal failure worsened (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Kidney failure (Renal and urinary disorders) | 1 (1) | 7 (7) | 2 (2)
Kidney function abnormal (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cellulitis of foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Gangrene (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Blood transfusion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gallbladder removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee surgery NOS (Surgical and medical procedures) | 0 (0) | 3 (3) | 0 (0)
Leg amputation (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1)
Open heart surgery (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension worsened (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Internal carotid aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemic stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)
Stroke (cerebrovascular accident) (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Stroke - Ischemic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unilateral Aflibercept- Monotherapy Group (N=116) | Unilateral Bevacizumab-First Group (N=112) | Bilateral Participants (N=42)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6) | 3 (3)
Anemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphangitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Heart block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral regurgitation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tricuspid regurgitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 0 (0)
Otitis media acute (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus poor control (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 1 (1)
Loss of control of blood sugar (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Worsening of diabetes (Endocrine disorders) | 7 (7) | 5 (5) | 2 (2)
Abnormal vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Anatomical narrow angle borderline glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anterior chamber cell (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Arcus senilis (Eye disorders) | 1 (1) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Blepharitis (eyelid irritation) (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 4 (4) | 7 (9) | 0 (0)
Blurry vision (Eye disorders) | 3 (4) | 2 (2) | 1 (1) — Affected (# Events): 1 (1) in Bevacizumab-First Group.
Borderline glaucoma (glaucoma suspect) (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Branch retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Burning eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 19 (19) | 7 (7) | 6 (13) — Affected (# Events): 6 (8) in Aflibercept-Monotherapy Group, 4 (5) in Bevacizumab-First Group.
Cataract cortical (Eye disorders) | 2 (2) | 3 (3) | 2 (4) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group, 2 (2) in Bevacizumab-First Group.
Central retinal vein occlusion (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Chemosis (conjunctival edema) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Choroidal nevus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Bevacizumab-First Group.
Cloudy vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Color vision change (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (3) | 2 (2) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group.
Contusion of orbital tissues (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Eye disorders) | 2 (2) | 1 (1) | 3 (4) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 2 (3) in Bevacizumab-First Group.
Corneal defect (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal endothelial disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Corneal epithelium defect (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal haze (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Corneal scar (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cortical spoking (Eye disorders) | 2 (2) | 2 (2) | 0 (0)
Cotton wool spots (Eye disorders) | 4 (4) | 3 (3) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Cupping of optic nerve (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cystoid macular edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic macular edema (Eye disorders) | 3 (4) | 5 (5) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Disc neovascularization (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Dry eye (Eye disorders) | 7 (7) | 2 (2) | 2 (4) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group, 2 (2) in Bevacizumab-First Group.
Dry eye syndrome (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 3 (3) | 1 (1) | 2 (2) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group.
Eye ache (Eye disorders) | 1 (2) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 2 (4) — Affected (# Events): 2 (3) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Eye pain (Eye disorders) | 6 (10) | 3 (3) | 3 (3) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye tearing (Eye disorders) | 1 (1) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Eyelid pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Flame-shaped hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 10 (13) | 9 (10) | 4 (7) — Affected (# Events): 3 (3) in Aflibercept-Monotherapy Group, 4 (4) in Bevacizumab-First Group.
Foreign body sensation in eyes (Eye disorders) | 4 (4) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Glaucoma (Eye disorders) | 1 (1) | 2 (2) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Hordeolum (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Hypertensive retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Incipient senile cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraretinal microvascular abnormalities (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iris neovascularization (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Iritis (anterior uveitis, iridocyclitis) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lattice degeneration of retina (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Lens disorder NOS (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Macular edema (Eye disorders) | 0 (0) | 0 (0) | 2 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Macular hole (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Macular ischemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Neovascular glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Nuclear sclerosis (Eye disorders) | 2 (2) | 2 (2) | 2 (3) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Ocular discomfort (Eye disorders) | 2 (2) | 1 (1) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Ocular hypertension (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Optic disc disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Bevacizumab-First Group.
Posterior capsule opacification (Eye disorders) | 3 (3) | 4 (5) | 2 (3) — Affected (# Events): 2 (2) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Posterior subcapsular cataract (Eye disorders) | 11 (13) | 3 (3) | 5 (9) — Affected (# Events): 4 (5) in Aflibercept-Monotherapy Group, 4 (4) in Bevacizumab-First Group.
Posterior vitreous detachment (Eye disorders) | 5 (5) | 7 (7) | 3 (3) — Affected (# Events): 3 (3) in Aflibercept-Monotherapy Group.
Preretinal hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Proliferative diabetic retinopathy (Eye disorders) | 2 (2) | 1 (1) | 1 (1) — Affected (# Events): 1 (1) in Bevacizumab-First Group.
Punctate epithelial erosion (Eye disorders) | 2 (2) | 1 (1) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Red eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal angiosclerosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1) | 1 (3) — Affected (# Events): 1 (2) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Retinal edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal exudates (Eye disorders) | 3 (3) | 6 (8) | 0 (0)
Retinal hemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal hole (Eye disorders) | 0 (0) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Retinal microaneurysms NOS (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Retinal pigment epitheliopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinoschisis (Eye disorders) | 0 (0) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Scleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Sensitivity to light (photophobia) (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Serous retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Silicone oil droplets (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Soreness in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Subconjunctival hemorrhage (Eye disorders) | 9 (19) | 10 (13) | 7 (27) — Affected (# Events): 6 (14) in Aflibercept-Monotherapy Group, 4 (13) in Bevacizumab-First Group.
Subconjunctival/conjunctival hemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Subretinal hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Bevacizumab-First Group.
Superficial punctate keratitis (Eye disorders) | 1 (1) | 5 (8) | 4 (7) — Affected (# Events): 4 (4) in Aflibercept-Monotherapy Group, 3 (3) in Bevacizumab-First Group.
Swollen eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Swollen eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Traction retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision abnormal (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 3 (3) | 4 (4) | 2 (3) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 2 (2) in Bevacizumab-First Group.
Visual acuity decreased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual disturbances (Eye disorders) | 0 (0) | 1 (1) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual flashes (Eye disorders) | 3 (3) | 2 (2) | 0 (0)
Vitreal cells (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreomacular traction syndrome (Eye disorders) | 0 (0) | 5 (5) | 0 (0)
Vitreous floater (Eye disorders) | 6 (6) | 2 (2) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Vitreous hemorrhage (Eye disorders) | 3 (3) | 4 (4) | 7 (11) — Affected (# Events): 4 (6) in Aflibercept-Monotherapy Group, 5 (5) in Bevacizumab-First Group.
Vitreous opacities (Eye disorders) | 1 (1) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Vitreous opacity (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group.
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (2) — Affected (# Events): 1 (1) in Aflibercept-Monotherapy Group, 1 (1) in Bevacizumab-First Group.
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acid reflux (oesophageal) (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Bloody stool (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Disease Crohns (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastro intestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocytic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (5) | 0 (0)
Reflux esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal bacterial overgrowth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach virus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3) | 3 (3)
Ache NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anasarca (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (3) | 2 (3) | 0 (0)
Chest pressure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dialysis access malfunction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (3) | 2 (2) | 1 (1)
Fever (General disorders) | 2 (4) | 1 (1) | 0 (0)
General Swelling (General disorders) | 3 (3) | 1 (1) | 2 (2)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Leg edema (General disorders) | 3 (3) | 1 (1) | 0 (0)
Localized superficial swelling, mass, or lump (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pedal edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of feet (General disorders) | 0 (0) | 2 (2) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 4 (4) | 1 (1) | 1 (1)
Abscess NOS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Enterococcus faecalis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foot infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fungal infection of nail (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infected toe (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 4 (4) | 2 (2)
MRSA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Septicemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Yeast infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 6 (9) | 1 (1)
Foot injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Knee injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Leg injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ligament tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spider bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0)
Angiogram (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine abnormal NOS (Investigations) | 0 (0) | 1 (1) | 0 (0)
Elevated liver enzymes (Investigations) | 0 (0) | 1 (1) | 0 (0)
Esophagogastroduodenoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Free prostate-specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
HbA1C increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Intraocular pressure increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
LDL cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation low (Investigations) | 1 (1) | 0 (0) | 0 (0)
Potassium high (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Testosterone low (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Fluid overload - fluid volume increased (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Folic acid deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesteremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2)
Water retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle injury (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Back discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Fractured ribs (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hand pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc bulging (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2)
Necrotizing fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in hip (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Painful feet (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Shoulder blade pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Shoulder fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sprains and strains of ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of knees (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
temporomandibular joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Consciousness loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 3 (3) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fainting (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head pressure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (2) | 2 (2)
Lumbar spinal stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory deficit (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Numbness generalized (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudotumor cerebri (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
VIth nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0)
Walking difficulty - Neurologic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Weakness left or right side (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Difficulty sleeping (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Bladder infection (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 4 (4) | 0 (0)
Chronic renal failure worsened (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (blood in urine) (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Kidney failure (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Kidney function abnormal (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Kidney infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Overactive bladder (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 6 (6) | 6 (7) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Enlarged prostate (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (8) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disease obstructive (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (7) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blister of foot and toe(s), without mention of infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Boil (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of foot (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Cellulitis of leg (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Congenital nevus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatochalasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Erythematous conditions (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Leg ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin bacterial infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin callus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)
Cataract extraction (Surgical and medical procedures) | 2 (2) | 2 (2) | 0 (0)
Debridement (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Knee surgery NOS (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Pacemaker insertion (cardiac) (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Root canal procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Claudication (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Embolism - blood clot (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 5 (5) | 5 (5)
Hypertension worsened (Vascular disorders) | 9 (10) | 3 (4) | 7 (8)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischemic attacks (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT03321513/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03321513/SAP_002.pdf
  • Informed Consent Form (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03321513/ICF_000.pdf